CLINICAL TRIAL: NCT07036367
Title: The Use of Sublingual Melatonin Premedication in Geriatric Cataract Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of clinical pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 33/2025
Record Dates: First submitted 2025-06-14; First posted 2025-06-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-06

CONDITIONS: Cataract Surgery Anesthesia
Keywords: Melatonin; Geriatric; Cataract Surgery; Premedication; Sedation; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin Group (Active Comparator): a 6 mg sublingual tablet of melatonin will be administered for all patients at 60 minutes before surgery.
  Interventions: Drug: Sublingual Melatonin
- Placebo Group (Placebo Comparator): the participants will be received a visually identical tablet containing inert ingredients at 60 minutes before surgery.
  Interventions: Drug: Sublingual Placebo

INTERVENTIONS:
Drug: Sublingual Melatonin — Participants in this group received 3 mg of sublingual melatonin, administered 60 minutes before cataract surgery. The melatonin was given in the form of a rapidly dissolving sublingual tablet to enhance bioavailability and ensure consistent preoperative absorption. The goal of the intervention was to reduce preoperative anxiety, improve sedation level, and stabilize hemodynamic parameters. The melatonin tablets were indistinguishable in appearance from the placebo and were prepared and dispensed by a pharmacy technician not involved in data collection or patient care
  Arms: Melatonin Group
Drug: Sublingual Placebo — Participants in this group received an identical-appearing sublingual placebo tablet containing inert ingredients, administered 60 minutes before cataract surgery. The placebo was visually indistinguishable from the melatonin tablets and was used to maintain double blinding in the trial. Tablets were prepared by the pharmacy team to ensure concealment and eliminate bias. This group was designed to serve as a control to evaluate the effectiveness of sublingual melatonin on anxiety and sedation levels in elderly patients
  Arms: Placebo Group

SUMMARY:
Cataract surgery is routinely performed with anesthesia care, whereas anesthesia care for other elective, low-risk, outpatient procedures is applied more selectively. We hypothesize that sublingual melatonin will provide superior anxiolysis and sedation while maintaining a high safety profile and minimizing hemodynamic disturbances.

DETAILED DESCRIPTION:
Prevalence of anesthesia care during cataract surgery compared with other low-risk procedures; association of anesthesia care with patient, clinician, and health system characteristics; and proportion of patients experiencing a significant anxiety and hemodynamic instability during cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 60 years

  * American Society of Anesthesiologists (ASA) physical status I-III
  * Scheduled for unilateral cataract surgery under local anesthesia
  * Ability to understand and complete study-related questionnaires

Exclusion Criteria:

* • Known allergy or hypersensitivity to melatonin

  * Chronic use of sedatives, hypnotics, or anxiolytics
  * History of sleep disorders or psychiatric illness
  * Visual or hearing impairment that would hinder communication
  * Emergency surgery or anticipated intraoperative complications

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
perioperative anxiety | at 30 and 60 minutes before procedure, with application of local anesthesia, 15 and 30 minutes after anesthesia.
  It will be assessed using the Visual Analog Scale (VAS) for anxiety (0-10 cm) upon arrival to the operating room.

CONTACTS AND LOCATIONS:
Overall Officials: Neveen A Kohaf, PhD, Principal Investigator — Al-Azhar University
Locations (2):
- Al-Azhar University, Cairo, Egypt, Egypt
- Al-Azhar University, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the principal investigator.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Wahane VD. A comparison of Gabapentin and melatonin for cataract surgery. Journal of Advanced Medical and Dental Sciences Research. 2017;5(8).